CLINICAL TRIAL: NCT04182152
Title: Bronchoscopic ICG Injection vs Percutaneous Hook-wire Techniques for Preoperative Lung Nodule Localization in Video-assisted Thoracoscopic Sublobar Resection: A Prospective and Randomized Trial
Brief Title: Bronchoscopic ICG Injection and Percutaneous Hook-wire Techniques for Preoperative Lung Nodule Localization in VATS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiayuan Sun (Other)
Responsible Party: Sponsor-Investigator, Jiayuan Sun, Director, Department of Endoscopy, Shanghai Chest Hospital, Shanghai Chest Hospital
Organization: Shanghai Chest Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SHCHE201905
Record Dates: First submitted 2019-11-26; First posted 2019-12-02 (Actual); Last update posted 2019-12-02 (Actual); Status verified 2019-11

CONDITIONS: Lung Cancer
Keywords: Electromagnetic navigation bronchoscopy (ENB); localization; Lung cancer; Video-associated thoracic surgery; Indocyanine green (ICG)
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bronchoscopic ICG localization (Experimental): The nodule will be located preoperatively by ENB-Guided bronchoscopic ICG injection; During the VATS operation, a near-infrared fluorescence thoracoscopy will be used to identify ICG distribution in the visceral pleura to guide an accurate surgical resection.
  Interventions: Device: Indocyanine green (ICG); Device: Electromagnetic navigation bronchoscopy
- percutaneous hook-wire localization (Active Comparator): The nodule will be located preoperatively by percutaneous placement of hook wire; During the VATS operation, the resection scope is determined by the location relationship between hook wire and the nodule under CT scan.
  Interventions: Device: Hook wire

INTERVENTIONS:
Device: Indocyanine green (ICG) — Indocyanine green (ICG) was diluted with saline to 0.5mg/mL, and injected 0.6mL/site.
  Arms: Bronchoscopic ICG localization
Device: Electromagnetic navigation bronchoscopy — Electromagnetic navigation bronchoscopy (ENB) allows physicians to access peripheral lung nodules with high accuracy and provides a working channel for ICG injection.
  Arms: Bronchoscopic ICG localization
Device: Hook wire — Hook wire is a puncture locating needle with a hook head that is about 1 cm in length and 30 cm metal wire behind. Through the puncture path planned based on CT scan, hook wire puncture percutaneously into the chest cavity to reach the lesion for localization.
  Arms: percutaneous hook-wire localization

SUMMARY:
The purpose of the study is to evaluate the efficacy and safety of transbronchial ICG and percutaneous hook-wire assisted Video-assisted thoracoscopic sublobar resection. In the control group, CT-guided percutaneous hook-wire preoperative localization will be used for surgical resection; In the experimental group, electromagnetic navigation bronchoscopy guided transbronchial ICG injection will be performed for localization before VATS.

DETAILED DESCRIPTION:
This is a single-center, prospective, randomized trial initiated by the investigator. Subjects with pulmonary nodules who will undergo Video-assisted thoracoscopic sublobar resection will be randomly divided into two groups. In the experimental group, before the VATS operation, transbronchial ICG injection will be guided by electromagnetic navigation bronchoscopy to locate the nodule. In the control group, the subject will undergo CT guided hook-wire placement for nodule localization before VATS. The study is expected to enroll 188 patients. Finally, the effectiveness and safety of the two methods will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Above 18 years old;
* With lung nodule diameter ≤2cm and distance from pleura ≥1cm, and VATS sublobar resection is arranged;
* Located difficultly by intraoperative visual inspection and palpation, a preoperative location is needed.

Exclusion Criteria:

* Cardiopulmonary function cannot tolerate general anesthesia, or other contraindications, such as uncorrectable coagulopathy;
* More than one pulmonary nodule requires preoperative localization;
* Subject underwent thoracic surgery in the past and was suspected of having severe chest adhesions;
* The nodule puncture path has bony structure block;
* Others conditions that the investigator considers not appropriate for this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Estimated)
Dates: Start 2019-11-05 (Actual); Primary Completion 2020-11-05 (Estimated); Study Completion 2020-12-05 (Estimated)

PRIMARY OUTCOMES:
Success rate of the localization procedure | On the 1 day of localization operation
  Calculated as follows: (number of successful targeting procedures/number of all localization procedures)*100
Success rate of the effective localization | On the 1 day of VATS operation
  Calculated as follows: [(number of successful targeting procedures-number of dislodgements or unrecognized in the operative field)/number of all localization procedures]*100
Success rate of VATS sublobar resection | On the 1 day of VATS completion
  Calculated as follows: (number of successful VATS procedures/number of all localization procedures)*100

SECONDARY OUTCOMES:
Safety endpoint | On the 1 day of VATS operation
  Complication rate of two localization methods, including pneumothorax, hemorrhage, etc.
Localization time | On the 1 day of localization operation
  The localization time of the control group was defined as the time from the first CT scan which set the path for percutaneous puncture, to the last CT scan which confirmed the hook wire located at the expected site.
  The localization time of the experimental group was defined as the time from the insertion of bronchoscope to the glottis, to the withdrawal of bronchoscope from the glottis after ICG injection.
Operation time of VATS sublobar resection | On the 1 day of VATS completion
  The operation time is defined as the time from the start of the skin incision to the completion of the suture of the skin.

CONTACTS AND LOCATIONS:
Overall Officials: Jiayuan Sun, MD, Principal Investigator — Shanghai Chest Hospital
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Altorki N, Shostak E. Localizing small nodules: Is it time for a randomized trial? J Thorac Cardiovasc Surg. 2017 Jun;153(6):1591. doi: 10.1016/j.jtcvs.2017.02.037. Epub 2017 Mar 8. No abstract available. PMID 28343689
- [Background] Park CH, Han K, Hur J, Lee SM, Lee JW, Hwang SH, Seo JS, Lee KH, Kwon W, Kim TH, Choi BW. Comparative Effectiveness and Safety of Preoperative Lung Localization for Pulmonary Nodules: A Systematic Review and Meta-analysis. Chest. 2017 Feb;151(2):316-328. doi: 10.1016/j.chest.2016.09.017. Epub 2016 Oct 4. PMID 27717643
- [Background] Zhang L, Wang L, Kadeer X, Zeyao L, Sun X, Sun W, She Y, Xie D, Li M, Zou L, Rocco G, Yang P, Chen C, Liu CC, Petersen RH, Ng CSH, Parrish S, Zhang YS, Giordano R, di Tommaso L; AME Thoracic Surgery Collaborative Group. Accuracy of a 3-Dimensionally Printed Navigational Template for Localizing Small Pulmonary Nodules: A Noninferiority Randomized Clinical Trial. JAMA Surg. 2019 Apr 1;154(4):295-303. doi: 10.1001/jamasurg.2018.4872. PMID 30586136
- [Background] Sun J, Mao X, Xie F, Han B, Chen H. Electromagnetic navigation bronchoscopy guided injection of methylene blue combined with hookwire for preoperative localization of small pulmonary lesions in thoracoscopic surgery. J Thorac Dis. 2015 Dec;7(12):E652-6. doi: 10.3978/j.issn.2072-1439.2015.12.24. PMID 26793384
- [Background] Sekine Y, Ko E, Oishi H, Miwa M. A simple and effective technique for identification of intersegmental planes by infrared thoracoscopy after transbronchial injection of indocyanine green. J Thorac Cardiovasc Surg. 2012 Jun;143(6):1330-5. doi: 10.1016/j.jtcvs.2012.01.079. Epub 2012 Feb 22. PMID 22361249
- [Background] Anayama T, Qiu J, Chan H, Nakajima T, Weersink R, Daly M, McConnell J, Waddell T, Keshavjee S, Jaffray D, Irish JC, Hirohashi K, Wada H, Orihashi K, Yasufuku K. Localization of pulmonary nodules using navigation bronchoscope and a near-infrared fluorescence thoracoscope. Ann Thorac Surg. 2015 Jan;99(1):224-30. doi: 10.1016/j.athoracsur.2014.07.050. Epub 2014 Nov 6. PMID 25442988
- [Background] Abbas A, Kadakia S, Ambur V, Muro K, Kaiser L. Intraoperative electromagnetic navigational bronchoscopic localization of small, deep, or subsolid pulmonary nodules. J Thorac Cardiovasc Surg. 2017 Jun;153(6):1581-1590. doi: 10.1016/j.jtcvs.2016.12.044. Epub 2017 Feb 7. PMID 28314525
- [Background] Hyun K, Park IK, Song JW, Park S, Kang CH, Kim YT. Electromagnetic navigation bronchoscopic dye marking for localization of small subsolid nodules: Retrospective observational study. Medicine (Baltimore). 2019 Mar;98(11):e14831. doi: 10.1097/MD.0000000000014831. PMID 30882669
- [Background] Anayama T, Hirohashi K, Miyazaki R, Okada H, Kawamoto N, Yamamoto M, Sato T, Orihashi K. Near-infrared dye marking for thoracoscopic resection of small-sized pulmonary nodules: comparison of percutaneous and bronchoscopic injection techniques. J Cardiothorac Surg. 2018 Jan 12;13(1):5. doi: 10.1186/s13019-018-0697-6. PMID 29329549